CLINICAL TRIAL: NCT07118670
Title: A 96-week, Single-arm Study to Evaluate the Efficacy and Safety of 8mg Aflibercept in Subjects With Proliferative Diabetic Retinopathy (PDR) Without Center-involved Diabetic Macular Edema (DME)
Brief Title: High Dose Eylea for Proliferative Diabetic Retinopathy Outcomes
Acronym: HERO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Edward Wood, MD (Other)
Collaborators: Greater Houston Retina Research (Other)
Responsible Party: Sponsor-Investigator, Edward Wood, MD, Principal Investigator, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe(HD)-DR-24143
Record Dates: First submitted 2025-07-29; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Proliferative Diabetic Retinopathy (PDR)
Keywords: HERO; PDR
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Subjects will receive 8mg aflibercept at week 0, 4, and 8. At week 8, subjects will enter a variable treatment and extension approach where they may be extended by 4-week intervals with no maximum interval between treatments until the end of study visit at week 96.
  Supplemental: Disease activity will be assessed at every 4-week visit and supplemental treatment with panretinal photocoagulation (PRP) as needed and/or intravitreal (IVT) 8mg aflibercept injections as determined by the regression patterns listed below.
  No regression: subjects will receive 8mg aflibercept and PRP every 4 weeks until they exhibit total regression, whereafter they may be re-extended.
  Partial regression: subjects will receive 8mg aflibercept every 8 weeks and not be extended until total regression is exhibited.
  Interventions: Drug: Aflibercept 8mg

INTERVENTIONS:
Drug: Aflibercept 8mg — Solution in Vial, intravitreal (IVT) injection
  Other Names: Eylea HD; 8 mg Aflibercept; Aflibercept High Dose VEGF Trap-Eye

SUMMARY:
The purpose of this Phase 4 study is to evaluate the safety of aflibercept 8mg in patients with proliferative diabetic retinopathy without center-involved diabetic macular edema.

DETAILED DESCRIPTION:
Subjects will be administered intravitreal aflibercept 8mg every 4 weeks, starting at week 0 for 8 weeks, then may be extended by 4-week intervals with no maximum between treatments with an end of study visit at week 96. At any visit, it will be determined if supplemental treatment is needed as determined by disease activity assessment until there is no regression of disease is noted and the extension intervals will begin again.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent
* Men or women > 18 years of age at the time of signing the Informed Consent Form
* Diagnosed with type 1 or type 2 diabetes mellitus
* BCVA ETDRS >/= 20/400 in the study eye
* Proliferative Diabetic Retinopathy as diagnosed via clinical examination and fluorescein angiography

Exclusion Criteria:

* Any known hypersensitivity to any of the components of aflibercept 8 mg injection
* Any known hypersensitivity to any contrast media (e.g., fluorescein), dilating eye drops, disinfectants (e.g., iodine), or any of the anesthetics and antimicrobial preparations used bye the site during the study
* Prior systemic anti-VEGF or IVT anti-VEGF treatment in the study eye within 3 months of enrollment. (i.e., 3-month wash-out period for anti-VEGF allowed)
* Any intra- or periocular corticosteroid treatment in the study eye within 3 months of baseline
* Any intraocular sustained-release treatment or implantable device
* Any gene therapy in the study eye
* SD-OCT central subfield thickness measurement of > 320 µm, in the study eye
* Evidence of ocular infection, in the study eye, at time of screening
* IOP > 25 mmHg in the study eye
* Any intraocular inflammation/ infection in either eye within 12 weeks (84 days) of the screening visit
* History of vitreoretinal surgery in the study eye
* Any prior Panretinal laser photocoagulation (PRP) in the study eye
* Current vitreous hemorrhage obscuring clear view of the macula in the study eye
* Presence of tractional retinal detachment and/or pre-retinal fibrosis causing retinal elevation/ thickening
* Cataract surgery in the study eye within 4 weeks prior to Screening/ Day 0
* Blood pressure > 180/100 mmHg systolic/ diastolic, while seated
* Pregnant or breastfeeding women
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening/ baseline; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly).

  * Contraception is not required for men with documented vasectomy

    * Postmenopausal women must be amenorrhoeic for at least 12 months in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint - DRSS step improvement | Baseline through weeks 48 and 96
  Proportion of eyes with ≥ 2 step improvement in diabetic retinopathy severity scale (DRSS), as assessed by the central reading center

SECONDARY OUTCOMES:
DRSS Step Improvement | Baseline to week 24 and 96
  Proportion of eyes with ≥ 2 step improvement in diabetic retinopathy severity scale (DRSS), as assessed by the central reading center
Mean change in BCVA | Baseline through weeks 24, 48, 72, and 96
  Evaluate the mean change in the best corrected visual acuity (BCVA)
Conversion from PDR to NPDR | Baseline to weeks 24, 48, 72, 96.
  Proportion of eyes converting from proliferative diabetic retinopathy (PDR) to non-proliferative diabetic retinopathy (NPDR)
DRSS Step Improvement | Baseline to weeks 24, 48, 72, 96
  Proportion of eyes with >= 3 step improvement in diabetic retinopathy severity scale (DRSS)
Retinal non-perfusion change | Baseline to weeks 24, 48, 72, 96.
  Mean change (quantitative area) in retinal vascular non-perfusion (RNP) based on ultrawide-field fluorescein angiography (UWFA)
Changes in visual function on HVF | Baseline to weeks 48, 96.
  Mean change in Humphrey visual field 30-2 total point score
CST change | Baseline to weeks 24, 48, 72, 96
  Mean change in CST
Number of supplemental treatments | Baseline through week 96
  Mean and median number of intravitreal (IVT) 8mg aflibercept injections (with and without intravitreal 8 mg aflibercept injections given for DME) as well as annualized injection frequencies
Worsening PDR | Baseline to week 96
  Mean time to development of worsening proliferative diabetic retinopathy associated event/s, including PDR-related vitrectomy, new or worsening preretinal or vitreous hemorrhage, retinal detachment, panretinal photocoagulation
CI-DME development | Baseline to week 96
  Mean time to development of central-involved DME (CI-DME)
AEs notated | Baseline to week 96
  Incidence and severity of ocular and systemic adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Edward Wood, MD, Principal Investigator — Retina Consultants of Texas

IPD SHARING:
Plan to Share IPD: No